CLINICAL TRIAL: NCT07271225
Title: Effectiveness and Safety of Auricular Acupuncture for Nausea and Vomiting Side Effects Induced by Anti-Tuberculosis Drugs in Pulmonary TB Patients
Brief Title: Safety and Efficacy of Ear Acupuncture for Antituberculosis Drug-Related Nausea and Vomiting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Kevin Supratman, MD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0215
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Intervention Model Description: The intervention group will receive press needle, while the control group will receive sham press needle
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding will be applied to participants and outcome assessors. Group allocation will not be disclosed to them to minimize assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Press Needle Group (Experimental): Press Needle
  Interventions: Device: Press Needle
- Sham Press Needle Group (Sham Comparator): Sham Press Needle
  Interventions: Device: Sham Press Needle

INTERVENTIONS:
Device: Press Needle — Press needle is performed once at bilateral MA-TF1 Shenmen, MA-AH-7 Sympathetic, and MA-IC6 Stomach using Press Needle (Pyonex® 0,17x0,9 mm). Standard aseptic procedures are followed. Participants continue their routine pharmacological anti-emetics treatment.
  Arms: Press Needle Group
Device: Sham Press Needle — Press needle is performed once at bilateral MA-TF1 Shenmen, MA-AH-7 Sympathetic, and MA-IC6 Stomach using Sham Press Needle. Standard aseptic procedures are followed. Participants continue their routine pharmacological anti-emetics treatment.
  Arms: Sham Press Needle Group

SUMMARY:
This study will look at whether press-needle ear acupuncture can help lower nausea and vomiting caused by antituberculosis medicines in people with pulmonary tuberculosis. Nausea and vomiting are common side effects of tuberculosis treatment, and they can make people stop taking their medicines

When treatment is stopped too early, tuberculosis may not be cured and may become resistant to medicines.

Participants in this study will have nausea and vomiting related to their tuberculosis treatment. They will be randomly assigned to one of two groups. One group will receive press-needle ear acupuncture. The other group will receive a placebo version that looks similar but does not stimulate acupuncture points

Researchers will check nausea and vomiting scores before treatment, during treatment, and after treatment to see whether press-needle acupuncture works better than placebo and whether it is safe. Press-needle acupuncture may help reduce nausea and vomiting by affecting nerves and lowering certain chemicals that trigger these symptoms, and it has minimal side effects

If this method is proven helpful and safe, it may give patients a comfortable and low-risk way to manage nausea and vomiting during tuberculosis treatment

ELIGIBILITY:
Inclusion Criteria:

* Participants are individuals diagnosed with drug-sensitive tuberculosis or drug-resistant tuberculosis receiving short-term treatment regimens (BPaL/BPaLM)
* Participants are aged 17 years or older.
* Participants experience nausea and vomiting after taking antituberculosis drugs.
* Participants are willing to comply with the study schedule until completion and provide written informed consent.

Exclusion Criteria:

* Presence of skin lesions at the site where press needles (PN) will be applied
* Participants who experience nausea and vomiting prior to antituberculosis treatment (including comorbidities that may cause nausea and vomiting, such as renal failure and liver disorders)
* Participants with drug-resistant tuberculosis (DR-TB) receiving long-term or individualized treatment regimens
* Participants with diabetes mellitus and a random blood glucose level > 200 mg/dL
* Participants with unstable hemodynamic status
* Participants who have received acupuncture therapy within the last 2 weeks
* Participants with coagulation disorders (platelet count < 50,000/µL)
* Participants with a history of hypersensitivity reactions to previous acupuncture treatment

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rhodes indeks of nausea, vomiting, and retching (RINVR) | Baseline, 1 day, 3 days, 7 days, 10 days, 14 days after intervention
  a validated patient-reported questionnaire used to measure the severity and impact of nausea, vomiting, and retching. It consists of eight items that evaluate the frequency, duration, and distress associated with these symptoms over a specific time period. Each item is scored using a Likert scale, and the total score reflects the overall symptom burden.

SECONDARY OUTCOMES:
Adverse Events Related to Intervention | 1 day, 3 days, 7 days, 10 days, 14 days after intervention
  Any adverse events occurring after the intervention, including infection, pain, or skin irritation at the insertion site, will be monitored and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- RSUP Persahabatan, Jakarta, Jakarta Timur, Indonesia

IPD SHARING:
Plan to Share IPD: No